CLINICAL TRIAL: NCT00498264
Title: Effectiveness of Physical Exercise on Decrease of Pain in Patients With Fibromyalgia:Randomized Clinical Trial
Brief Title: Effectiveness of Physical Exercise in Women With Fibromyalgia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of São Paulo (Other)
Collaborators: University of Santo Amaro (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AHK12121977
Record Dates: First submitted 2007-07-09; First posted 2007-07-10 (Estimated); Last update posted 2007-07-10 (Estimated); Status verified 2007-06

CONDITIONS: Fibromyalgia
Keywords: Exercise; Rehabilitation; Strength exercise; Aerobic exercise; Pain
MeSH Terms: conditions — Fibromyalgia; Motor Activity; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: walking program, resistance muscular exercise

SUMMARY:
Fibromyalgia (FMS) is a syndrome expressed by chronic widespread body pain which leads to reduced physical function and frequent use of health care services. Exercise training is commonly recommended as a treatment.

The purpose of this study is to determine whether a supervised resistance muscular exercise (RME) and walking program (WP) are effective in the treatment of FMS on decrease of pain.

The practical of the RME reduces the pain of participants with FMS.

DETAILED DESCRIPTION:
This study will evaluate and compare the effectiveness of a supervised resistance muscular exercise (RME) , walking program (WP)and control group (just observation) in women with FMS during 16 weeks, on decrease of pain.

Participants will undergo an assessment including medical some questionnaires to assess their FMS symptoms at baseline, after 8 weeks, 16 weeks and 28 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Criteria diagnosis according ACR 1990
* Wash-out of medication specific for fibromyalgia for 1 month
* Only paracetamol 750mg will be allowed during the period of study.

Exclusion Criteria:

* Alterations that against indicate the practical one of physical activity evaluated previously in clinical and rheumatology evaluation

Ages: 35 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2005-01; Study Completion 2007-10 (Estimated)

PRIMARY OUTCOMES:
Decrease of pain and use of specific medicine for fibromyalgia | 16 weeks

SECONDARY OUTCOMES:
Improvement on phsysical function assessment throughout of 6 minute walk test and specific questionnaire: FIQ (Fibromyalgia Impact questionnarie) and SF-36 (Quality of life) | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Andrea H Kayo, PT, Principal Investigator — Federal University of São Paulo
Locations (1):
- University of Santo Amaro - Ambulatory of Special Conditions, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Kayo AH, Peccin MS, Sanches CM, Trevisani VF. Effectiveness of physical activity in reducing pain in patients with fibromyalgia: a blinded randomized clinical trial. Rheumatol Int. 2012 Aug;32(8):2285-92. doi: 10.1007/s00296-011-1958-z. Epub 2011 May 19. PMID 21594719